CLINICAL TRIAL: NCT00691600
Title: Phase 3 Study Comparing Bactrim to Placebo in the Management of Abscesses < 5cm in the Pediatric Population.
Brief Title: Management of Skin and Soft Tissue Abscesses in Pediatric Patients After Incision and Drainage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Andrea Cruz, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-18758
Record Dates: First submitted 2007-12-28; First posted 2008-06-05 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Abscess
Keywords: abscess; Abscesses in the pediatric emergency population
MeSH Terms: conditions — Abscess | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral trimethoprim/sulfamethoxazole (Active Comparator): subjects with abscesses less than 5cm will be randomized to either study med or placebo
  Interventions: Drug: oral trimethoprim/sulfamethoxazole
- placebo (Placebo Comparator): Placebo after incision and drainage of abscess less than 5 cm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral trimethoprim/sulfamethoxazole — 80 mg caps or 8 mg/ml suspension every 12 hours for 10 days
  Other Names: TMP/SMX
  Arms: oral trimethoprim/sulfamethoxazole
Drug: Placebo — Placebo caps or suspension every 12 hours for 10 days
  Other Names: Placebo caps
  Arms: placebo

SUMMARY:
The purpose of the study is to compare rates of cure of abscesses with and without antibiotic treatment after incision and drainage. The purpose of this study is to compare successful rates of cure of abscesses less than 5 cm with antibiotic (oral TMP/SMX) versus non-antibiotic treatment after incision and drainage.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of antibiotic treatment versus placebo after incision and drainage of skin and soft tissue abscesses less than 5 cm in pediatric patients. Eligible patients whose parents/guardians consented them to enrollment were randomized to receive one of two interventions: oral trimethoprim/sulfamethoxazole (TMP/SMX) or placebo after incision and drainage. Every attempt was made to make the placebo capsules and suspensions appear in all aspects like the true drug (was done by the investigational pharmacy department at our institution). Equal numbers of subjects were randomized at the outset to both study groups. Randomization, also done by our investigational pharmacy department, was done in blocks of 20. Patients were followed up in our emergency center at 24 to 48 hours to have any packing removed and to have their clinical/wound status assessed. They were not charged for this visit, and their valet parking was validated. If an individual patient, or an individual patient's wound, was felt to be not improving adequately, that patient was started on formal antibiotic therapy at the treating attending physician's discretion.

Primary outcome:

1. Abscess resolution by parental report 7-10 days after incision and drainage

Secondary outcomes:

1. Admission to the hospital because of worsening infection
2. Receipt of antibiotics (placebo arm) or change in antibiotics (antibiotic arm)

ELIGIBILITY:
Inclusion Criteria:

1.) Abscess < 5 cm (< 5 cm of induration and fluctuance) requiring incision and drainage 2.) Age > 90 days and < 18 years 3.) Abscess on the trunk, scalp, extremities, or axillae

Exclusion Criteria:

1. Multiple abscesses
2. Abscess located on the hands, face, or perineum
3. Abscess as a result of a bite wound
4. Immunocompromised patient - i.e., diabetes, sickle cell, chronic steroid therapy (> 10 days), etc.
5. Previously failed 48 hours or greater therapy on any antibiotic regimen 6.) Drug allergy to TMP/SMX

7.) Fever > or = 102.2 degrees Fahrenheit in the previous 24 hours 8.) Systemic symptoms on presentation - i.e., nausea , vomiting, persistent tachycardia, hypotension, diaphoresis, etc.

9.) Signs /symptoms of another infection or illness - i.e., influenza, croup, etc.

Ages: 90 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cruz, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotic Arm: subjects with abscesses less than 5cm will be randomized to oral trimethoprim/sulfamethoxazole: 80 mg caps or 8 mg/ml suspension every 12 hours for 10 days
- Placebo Arm: Patients with abscesses < 5cm randomized to placebo tablets or suspension twice a day for 10 days
Period: Overall Study
Arm/Group | Antibiotic Arm | Placebo Arm
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat
Groups:
- Oral Trimethoprim/Sulfamethoxazole: subjects with abscesses less than 5cm will be randomized to study medication, oral trimethoprim/sulfamethoxazole:
  80 mg caps or 8 mg/ml suspension every 12 hours for 10 days
- Placebo After Incision and Drainage: Patients with abscesses less than 5cm will be randomized to receive placebo.
  Placebo: Placebo capsules every 12 hours for 10 days
- Total: Total of all reporting groups
Arm/Group | Oral Trimethoprim/Sulfamethoxazole | Placebo After Incision and Drainage | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 11 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abscess Resolution
Description: Outcomes will be measured by resolution of size, tenderness, and induration with erythema by parental report 7 - 10 days after initial visit to the Emergency Center
Time Frame: 10 days
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Groups:
- Antibiotic Arm: oral trimethoprim/sulfamethoxazole: 80 mg caps or 8 mg/ml suspension every 12 hours for 10 days
- Placebo Arm: Receipt of placebo in either capsule or suspension formulation twice daily for 10 days
Arm/Group | Antibiotic Arm | Placebo Arm
Number analyzed (Participants) | 12 | 11
Participants | 11 | 9

2. Secondary Outcome: Number of Participants Requiring Admission for Failure of Abscess Resolution
Description: Percentage of patients requiring admission to Texas Children's or another hospital within 10 days of incision and drainage
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic Arm | Placebo Arm
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Requiring New or Modified Antibiotics for Failure of Abscess to Resolve
Description: For the antibiotic arm, we determined if the child was prescribed a different antibiotic.
  For the placebo arm, we determined if the child received a prescription for an antibiotic at a subsequent visit (e.g., in the emergency department, by their pediatrician, etc) within 10 days of incision and drainage
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic Arm | Placebo Arm
Number analyzed (Participants) | 12 | 11
Participants | 1 | 2

ADVERSE EVENTS:
Groups:
- Antibiotic Arm: subjects with abscesses less than 5cm who received oral trimethoprim/sulfamethoxazole: 80 mg caps or 8 mg/ml suspension every 12 hours for 10 days
- Placebo Arm: subjects with abscesses less than 5cm who received placebo capsules or suspension every 12 hours for 10 days
Arm/Group | Antibiotic Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No